CLINICAL TRIAL: NCT01747291
Title: Atypical Femur Fracture Ontario Cohort Registry
Brief Title: Atypical Fracture Cohort Study
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0532
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Atypical Femur Fracture; Atypical Subtrochanteric Fracture; Osteoporosis With AFf

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atypical femur fracture cohort

SUMMARY:
Osteoporosis is a disease characterized by increased bone fragility and deteriorating bone micro-architecture. The main consequence of osteoporosis is low-trauma fractures, most often of the hip, spine and wrist. Recently, another type of low-trauma fracture, atypical femur fractures (AFFs), have received much attention. Little is known of the cause of these debilitating fractures; however, they have been associated with long term bisphosphonate use. What we currently know about AFFs is based on case reports or small case series, or studies using administrative databases or secondary analyses of bisphosphonate trials. While these reports provide some preliminary information on the relationship between long term bisphosphonate exposure and AFFs, detailed clinical data are absent. As we have established a network of specialists across southern Ontario our group is in a position to collect meaningful information on a larger group of patients who have experienced these debilitating fractures into a centralized AFF registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 20;
* Patients who have experienced an incomplete AFF that satisfies the diagnostic criteria as set forth by the American Society of Bone and mineral Research (ASBMR) International Task Force on AFFs or a low (or no) trauma fracture that mimics the features described above at other sites.

Exclusion Criteria:

* Peri-prosthetic fractures;
* High trauma fractures;
* Pathological fractures secondary to metastases or metabolic bone diseases other than osteoporosis.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary or tertiary care clinic patients who have experienced an atypical fracture at any point in the past will be eligible for this observational study. Low trauma fractures are defined as fractures sustained with minimal force, such as a fall from standing height.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-06; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prospectively identify and diagnose atypical fracture patients in Ontario | baseline
  The objective of this exploratory study is to identify and diagnose AFF patients

SECONDARY OUTCOMES:
Examine risk factors and predictors for AFFs | baseline
  This exploratory study will examine risk factors and predictors for AFFs

OTHER OUTCOMES:
Examine how AFFs affect quality of life, functional recovery and health outcomes. | baseline and every 6-12 months
  This exploratory study will examine how AFFs affect quality of life, functional recovery and health outcomes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Angela m Cheung, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - University Health Network, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario